CLINICAL TRIAL: NCT01948583
Title: Humectant Activity of a New Formulation of Gynomunal® Vaginalgel: Crossover Test Use Versus Previous Formula
Brief Title: Humectant Activity of a New Formulation of Gynomunal® Vaginalgel
Acronym: GYNOMUNAL®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Dermatologist, Derming SRL
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E0513
Record Dates: First submitted 2013-09-06; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Vaginal Dryness; Menopause
Keywords: vaginal dryness; hyaluronic acid; menopause
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: vaginal gel new formulation (Active Comparator): Application once a day at evening during the first study week of the vaginal gel new formulation (hyaluronic acid).
  One week of wash-out (second week). Application once a day at evening during the third study week of the vaginal gel on the market (hyaluronic acid).
  Interventions: Drug: Hyaluronic Acid
- Arm II: vaginal gel on the market (Active Comparator): Application once a day at evening during the first study week of the vaginal gel on the market (hyaluronic acid).
  One week of wash-out (second week). Application once a day at evening during the third study week of the vaginal new formulation (hyluronic acid).
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Hyaluronic Acid — Arm I: new formulation applied for the first week, formulation on the marked applied for the third week (second week - wash out period) Arm II: formulation on the marked applied for the first week, new formulation applied for the third week (second week - wash out period)
  Other Names: Gynomunal® Vaginalgel (GYNOMUNAL®)

SUMMARY:
Aim of the study is to evaluate the humectant activity and the local tolerability of a new formulation of Gynomunal® vaginalgel in menopausal women (menopause since at least 2 years) with referred vaginal dryness

DETAILED DESCRIPTION:
Randomized, controlled, crossover clinical study; the subjects will use both formulations with an interval of 1 week (wash out period), in reversed sequence according to the treatment arm assigned at each subject during the basal visit.

Both tested products will be applied in the vagina, using the dedicated applicator, once a day, preferably at bedtime. To investigate the activity of the products under study, 4 visits will be performed: a baseline visit (T0), a visit at the end of the first week-treatment (T1), a visit at the end of the wash out period (T2) and a final visit at the end of the second week-treatment (T3).

Volunteers will be asked to follow their normal life and sexual habits, except for not having sexual intercourse 48 hours prior to each examination.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian healthy female subjects,
* complaining vaginal dryness,
* women in menopause since at least 2 years; the starting period of menopause being defined as the date when the last menstruation or metrorragia linked to hormonal unbalance took place,
* women who agree not to start a replacement therapy during the whole duration of the study,
* women who do not present any active cutaneous pathology of external and internal genitalia,
* women who did not receive any drug or cosmetic treatment on their genitalia during the 2 months preceding the trial,
* women who did not apply vaginal products within at least 1 month before the inclusion in the study,
* women who accept to use only the products authorised by the protocol,
* women who accept not to undertake any treatment for internal and external genitalia during the trial,
* women who did not use, phytoestrogenes based products on treated areas less than 4 weeks before inclusion time,
* women accepting to sign the Informed consent form,
* women able to read the material dedicated to volunteers, to abide by the rules of the protocol and ready to accept its constraints

Exclusion Criteria:

* Volunteers not fulfilling inclusion criteria,
* severe symptoms of vaginal dryness, associated with mucosal signs
* history of intolerance to a vaginal product,
* concomitant participation to another trial,
* refusal to sign the Informed Consent form,
* known allergy to one or several ingredients of the product on trial,
* change in the normal habits in the last 3 months,
* participation in a similar study during the previous 3 months,
* whose insufficient adhesion to the study protocol is foreseeable
* women who start a replacement therapy during the trial
* women who experience during the study the occurrence of any foreseeable risk to use daily the product on trial.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Vaginal Humidity determination | 2 weeks

SECONDARY OUTCOMES:
Tolerability assessment | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Physician, Principal Investigator — Derming SRL
Locations (1):
- DermIng S.r.l, Monza, MB, Italy